CLINICAL TRIAL: NCT05049187
Title: Characterization and Durability of COVID-19 Vaccine Induced Immune Responses in Healthcare/Frontline Workers
Status: Completed | Type: Observational
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: National Institute of Epidemiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021 007
Record Dates: First submitted 2021-09-17; First posted 2021-09-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 COVISHIELD: Participants will receive one dose of COVID-19 vaccine (Covishield) at baseline and one second dose after 28 days (Window period of +3 days) intra muscularly.
- Group 2 COVAXIN: Participants will receive one dose of COVID-19 vaccine (Covaxin) at baseline and one second dose after 28 days (Window period of +3 days) intra muscularly.

SUMMARY:
Rationale: Early in the covid-19 pandemic, it was unclear whether and how individuals and populations would develop protective and enduring immunity against SARS-CoV-2, either after infection or vaccination. It is still not clear what role might immune cellular responses play in the development of immunity to SARS-CoV-2 infection and what are the implications for vaccines? As T cells recognise and respond to viral antigens they produce many protective reactions and effector molecules. One such molecule is the cytokine interferon γ, secreted by CD4+ and CD8+ T cells and their memory cells. This can be measured means of documenting specific T cell responses to viral antigens. Published studies offered a strong evidence that T cell immune responses are sustained, even in the face of declining or undetectable antibodies, implying that some immunity persists. The evidence from new studies, interim results from phase III vaccine trials, and previous data from phase I and phase II trials support the notion that memory T cell responses to the vaccines, along with B cell antibody responses, should provide good and possibly enduring immunity to SARS-Cov-2. We propose to describe and characterize the humoral, innate and long-term adaptive immune responses and the neutralization potential generated by COVID-19 vaccination (Covaxin, Covishield) among healthcare and frontline workers.

DETAILED DESCRIPTION:
Study objectives i. To estimate the neutralizing antibodies titre against SARS CoV-2 by vaccine type.

ii. To estimate the proportion of vaccine recipients developing effective antibody response for SARS-CoV-2 specific IgG, IgM, and total IgE and IgA antibodies pre- and post-COVID-19 vaccination on day zero, day 28, month 2, 3, 6, 12, 18 and 24 by vaccine type.

iii. To identify and characterize the immune biomarkers for long term innate and adaptive immune response by vaccine type.

iv. To estimate the ratio of immune biomarker levels between pre- and post- COVID-19 vaccination at days 28, month 2, 3, 6, 12, 18 and 24 by vaccine type

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years
* Should have been vaccinated with either Covaxin or Covishield
* Willing to provide written informed consent

Exclusion Criteria:

* Participants will be ineligible if they are not vaccinated for either Covaxin or Covishield vaccine
* Not willing to provide written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthcare/frontline workers working in the ICMR-NIRT and ICMR-NIE aged 18 to 60 years
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Antibody titers | 2 years
  IgM and IgG SARS-Cov2 specific antibody titres and IgA and IgE (total)
Ratio of immune biomarker production | 2 years
  The ratio of immune biomarkers production between pre and post COVID-19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: PAVAN Kumar, PhD, Principal Investigator — National Institute for Research in Tuberculosis; BANUREKHA V V, MBBS, MPH, Principal Investigator — National Institute for Research in Tuberculosis
Locations (1):
- National Institute for Research in Tuberculosis, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No